CLINICAL TRIAL: NCT01600651
Title: Effects Of A Recruitment Maneuver On Plasma Levels of sRAGE, The Soluble Form of The Receptor For Advanced Glycation End Products, In Patients With Diffuse Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Diffuse Acute Respiratory Distress Syndrome (ARDS), Recruitment Maneuver, and sRAGE (DAMAGE Study)
Acronym: DAMAGE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CHU-0119
Record Dates: First submitted 2012-04-24; First posted 2012-05-17 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-10

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Receptor for advanced glycation end products (RAGE); Soluble RAGE (sRAGE); Recruitment Maneuver; Acute respiratory distress syndrome (ARDS); Alveolar epithelium; Electrical Impedance Tomography; Mechanical ventilation; Intensive Care Unit (ICU)
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Recruitment maneuver (RM) sham group (Sham Comparator): when recruitment maneuver sequence precedes a sham evaluation period
  Interventions: Other: Recruitment Maneuver (RM) sham group
- Sham Recruitment (RM) maneuver group (Sham Comparator): a group in which patients receive a sham sequence before the RM sequence
  Interventions: Other: Sham recruitment maneuver (RM) group

INTERVENTIONS:
Other: Recruitment Maneuver (RM) sham group — It 's when RM sequence precedes a shame evaluation period
  Arms: Recruitment maneuver (RM) sham group
Other: Sham recruitment maneuver (RM) group — Group in which patients receive a sham sequence before the RM sequence
  Arms: Sham Recruitment (RM) maneuver group

SUMMARY:
RAGE, the receptor for advanced glycation end products, is a novel marker of alveolar epithelial type I cell injury, and soluble RAGE (sRAGE) is elevated in the plasma and in the pulmonary edema fluid from patients with ALI/ARDS. Few data are available about the influence of ventilatory interventions on levels of sRAGE in the setting of ALI/ARDS. The purpose of this prospective monocentric randomized controlled cross-over study is to describe the effects of a recruitment maneuver (RM) on plasma sRAGE levels during diffuse ARDS.

DETAILED DESCRIPTION:
BACKGROUND:

The receptor for advanced glycation end products (RAGE) is now identified as a marker of alveolar type I cell injury. RAGE is a member of the immunoglobulin superfamily that acts as a multiligand receptor and is involved in propagating inflammatory responses. While the precise function of RAGE remains unclear, the elevated levels of RAGE, and its soluble isoform sRAGE, correlate with severity of ALI/ARDS in human and animal studies, and higher sRAGE levels could reflect impaired alveolar fluid clearance. Lung morphology, as assessed by loss of aeration distribution patterns on computed tomography (CT) scan, predicts the response to recruitment maneuvers in patients with ARDS: patients presenting with nonfocal (diffuse) lung morphology are more likely to respond to a RM, resulting in an increase in arterial oxygenation, net alveolar fluid clearance, and significant alveolar recruitment as revealed by pressure-volume curve analysis.

DESIGN NARRATIVE:

The purpose of this prospective, randomized and controlled, cross-over study is to compare the effects of a RM on plasma sRAGE levels (measured 5 minutes before, 5 minutes, 30 minutes, 1 hour, 4 hours and 6 hours after the RM) and plasma sRAGE levels measured during a "sham" or "control" sequence, in patients with diffuse ARDS.

Mechanically ventilated ICU patients with ARDS criteria (based on the 1994 American-European Consensus Conference definition for ARDS) and nonfocal CT scan lung morphology will be included within 24 hours of disease onset. Then, patients will be randomized into 2 groups: a "RM-SHAM" group when RM sequence precedes a sham evaluation period, and a "SHAM-RM" group, in which patients receive a sham sequence before the RM sequence. Patients will receive protective ventilation, as recommended, before, during and after evaluation periods. RM consists of the application of 40 cmH20 airway pressure for 40 seconds.

Blood will be sampled from an indwelling arterial catheter, in order to analyze arterial blood gases and sRAGE levels, 5 minutes before the RM (or a 40 second-long sham period), 5 minutes, 30 minutes, 1 hour, 4 hours and 6 hours after the RM (or a 40 second-long sham period). Electric impedance tomography will be evaluated 5 minutes before and 1 hour after the RM.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients under mechanical ventilation
* Patients within the first 24 hours after onset of ARDS according to the 1994 American-European Consensus Conference (AECC)
* PaO2/FiO2 ratio < 200 with external PEEP >5 cmH2O
* "Nonfocal" loss of aeration based on CT scan lung morphology analysis, as defined by the "CT scan ARDS study group" criteria

Exclusion Criteria:

* Pregnancy
* Acute exacerbation of diabetes
* Dialysis for end-stage kidney disease
* Alzheimer's disease
* Amyloidosis
* Evolutive neoplastic lesion
* Known or suspected history of allergy to cisatracurium
* Chronic respiratory disease requiring long term oxygen therapy or long term ventilation
* Confirmed or suspected elevated intracranial pressure
* Confirmed or suspected bronchopleural fistula, pneumothorax
* Persistent hemodynamic instability despite appropriate resuscitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Plasma sRAGE | 1 hour after the RM

SECONDARY OUTCOMES:
Plasma sRAGE in responders and non-responders to RM | 5 minutes before, then 5 minutes, 30 minutes, 4 hours and 6 hours after RM
Kinetics of sRAGE after RM | 5 minutes before, and 5 minutes, 30 minutes, 1 hour, 4 hours and 6 hours after RM and after a sham period
Predictive value of baseline sRAGE on the response to RM | 5 minutes before, and 5 minutes, 30 minutes, 1 hour, 4 hours and 6 hours after RM
Correlation of plasma sRAGE and response to RM with lung aeration | 5 minutes before, and 5 minutes, 30 minutes, 1 hour, 4 hours and 6 hours after RM or sham period
Risk of RM-related pulmonary bacterial translocation | 5 minutes before and 30 minutes after RM

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Jabaudon M, Hamroun N, Roszyk L, Guerin R, Bazin JE, Sapin V, Pereira B, Constantin JM. Effects of a recruitment maneuver on plasma levels of soluble RAGE in patients with diffuse acute respiratory distress syndrome: a prospective randomized crossover study. Intensive Care Med. 2015 May;41(5):846-55. doi: 10.1007/s00134-015-3726-0. Epub 2015 Mar 20. PMID 25792206